CLINICAL TRIAL: NCT02596113
Title: Νew Molecular Biomarkers for the Prevention and Early Detection of Precancerous or Cancerous Colorectal Lesions During Screening for Colorectal Cancer
Brief Title: Prevention and Early Detection Biomarkers of Adenomas and CRC Lesions During CRC Screening
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Director Gastroenterology, Evangelismos Hospital
Other Study IDs: galanopoulosm
Record Dates: First submitted 2015-10-03; First posted 2015-11-04 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; genes involved in carcinogenesis of the colon; screening colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood serum and colonic polyps tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- No pathological findings: blood and biopsy samples from normal colon mucosa
- >1 cm adenomatous polys: blood and biopsy samples from the polyp
- Colorectal cancer: blood (plasma) and biopsy samples from colorectal cancer

SUMMARY:
The investigators designed a prospective study to evaluate the predictive ability of detection of mutations in genes involved in carcinogenesis of the colon (eg hMLH1, K-Ras, B-Raf, ccfDNA) in a sample of Greek population presents for conducting colonoscopy in the context of screening under international CRC prevention instructions. This investigation will be carried out in individuals in normal risk in order to study specific mutations (in blood and tissue) to draw reliable conclusions about whether we can detect (with greater sensitivity and specificity) patients with precancerous lesions or CRC with a simple blood test thereby reducing the cost and side effects of repeated endoscopic procedures.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most frequent cancer worldwide with a prevalence of 1.5 million people / year and is the second cause of death from cancer (650 000 deaths per year) for both genders after lung cancer.

In Greece it is estimated that about 3000 people are infected annually by the CRC. Risk factors for the emergence of CRC are: old age, positive family history of cancer and colon polyps, diet poor in fiber and rich in high-calorie fats and foods, sedentary lifestyle and lack of exercise from everyday life. Additionally, obesity, smoking, alcohol consumption in large quantities, diabetes, inflammatory conditions of the intestine such as ulcerative colitis and Crohn's Crohn, and some inherited disorders affecting colon are factors that increase the risk for the CRC.

It is a silent and insidious disease since most patients do not present symptoms in the early stages (such as bleeding, abdominal pain), resulting in diagnosis in a non-curable phase. This makes it clear that survival depends on the stage of disease at time of diagnosis. For example a patient with cancer Dukes' stage A, 5-year survival is about 93% whereas stage C, is about 47%. Based on the above it is clear that early detection of precancerous colorectal lesions is the cornerstone for the optimal treatment of this disease.

The CRC is an ideally disease to implement mass screening in general population as it follows a specific development process that lasts 7-12 years, leading to transformation of normal epithelium to adenoma and eventually carcinoma.

There are multiple options available for CRC detection involving the detection of blood in fecal test (or microscopic examination of fecal hemoglobin), the flexible sigmoidoscopy and colonoscopy. Each of these has advantages and disadvantages. Specifically, the microscopic examination of fecal hemoglobin although reduces mortality by 16% by CRC nevertheless exhibits low sensitivity to detect polyps and cancerous lesions in the distal colon and small specificity thus be, in economic terms, negative test to be used in mass screening. Regarding the flexible sigmoidoscopy, this is a test clearly faster and safer than colonoscopy but with small percentage of patient compliance, efficacy clear depended on the quality of bowel preparation and most importantly, it can not see the whole intestine. Computed tomographic colonography is another method of finding new precancerous lesions but because of the short diagnostic accuracy compared to the colonoscopy and radiation, is not recommended for mass screening.

A colonoscopy is the best method for the diagnosis of polyps and CRC to date, and also prevents the CRC by detecting adenomatous polyps and through polypectomy. It allows the inspection of the entire lumen of the colon resulting in both distal and proximal lesions to be discovered. He has the greatest sensitivity by all methods in the detection of the CRC. The disadvantages of this method is the cost, bowel perforation and bleeding risks (especially after polypectomy), the difficulty in the preparation of patients using laxatives liquid, the need for sedation during the procedure, low levels of compliance and patient intolerance .

It becomes necessary to identify simpler, less invasive and more affordable methods of finding precancerous lesions for sporadic type of CRC. One such method is the use of potential biomarkers (i.e. objectively measurable indicators of a normal or abnormal process) using a sample of blood (plasma) of the person in order to find mutations or epigenetic changes in known genes that have been implicated to participate in the process of carcinogenesis of CRC.

More specific, there are at least three main paths that lead to carcinogenesis of colorectal lesions: the way of chromosomal instability (CIN), the path of microsatellite instability (MSI) and finally the path of methylated phenotype of the islands of cytosine-phosphate-guanine (CpG island) known as CpG Island Methylation Pathway (CIMP). After long-term studies, it has been found that in every path there is a participation of genes through their mutations and/or their epigenetic changes.

For example the path of chromosomal abnormality gathers the point mutations of some oncogenes and tumor suppressing genes such as APC, KRAS, BRAF, SMAD 4, and TP53.

The route of microsatellite instability, which is a result of the malfunctioning of the DNA repair genes (DNA mismatch repair genes -MMR), leads to multiple mutations and it is the cause of 15% of sporadic type of CRC by an abnormal epigenetic methylation of the MLH1gene. Eventually, the third path, CIMP, consists of two subtypes: the first is associated with mutations in the BRAF gene, known as CIMP-High, and the second associated with mutations in the KRAS gene, known as, CIMP-Low.

Additionally, the presence of circulating nucleic acids (circulating cell-free DNA) in the blood circulation in cancer patients has led to the belief that these nucleic acids derived from cancerous cells and therefore may be used in the early detection of precancerous or cancerous colorectal lesions.

Therefore it is becoming increasingly strong need to find new biomarkers that will lead us with lower costs and safety, closer to precancerous colon lesions, treating one of the most important health problems of our century.

Based on the above, we designed a prospective study to evaluate the predictive ability of detection of mutations in genes involved in carcinogenesis of the colon (eg hMLH1, K-Ras, B-Raf, ccfDNA) in a sample of Greek population presents for conducting colonoscopy in the context of screening under international CRC prevention instructions. This investigation will be carried out in individuals in normal risk in order to study specific mutations (in blood and tissue) to draw reliable conclusions about whether we can detect (with greater sensitivity and specificity) patients with precancerous lesions or CRC with a simple blood test thereby reducing the cost and side effects of repeated endoscopic procedures.

The sample to be studied will consist of approximately 90-100 individuals in normal risk for developing CRC aged 50-75 years, will undergo preventive colonoscopy for polyps and CRC detection. Participants will be divided into three groups of patients according to the findings during endoscopy: those without pathological findings, those with polyps between 1 to 3 centimeters diameter and adenomatous elements in pathology examination and finally those with colorectal cancer. From all these three populations, samples would be collected from peripheral blood (plasma) and colon tissue biopsy (normal or abnormal, respectively) in order to find a possible common mutations of some genes involved in the pathogenesis of the CRC in these 3 groups [e.g. in KRAS12, 13, 61, BRAF (V600E), ccfDNA some point mutations in hMLH1]. The samples of blood and tissue will be placed in a blood bottle with a specific anticoagulant and preservative (RNA latter) and subsequently stored at -20 degrees for maintenance. The genome analysis of potential mutations will be done by specific commercial DNA kit and specific PCR techniques. Then according to the results, it will be carried out a try to present statistically significant elements compatible or not with the original purpose of the investigation.

The effectiveness of the screening program depends on the accuracy and acceptability of the method used for detecting a pathological condition. An ideal screening test should have high compliance, high sensitivity and specificity, to be minimally invasive and cost-efficient. Because of the limitations of existing colon cancer screening methods there is a growing need to find new diagnostic methods for precancerous lesions and one of them are the molecular biomarkers that will be valuable tools in our arsenal to a safer approach to healthy subjects who are at high risk for CRC.

ELIGIBILITY:
Inclusion Criteria:

* normal risk for developing CRC aged 50-75 years who undergo preventive colonoscopy for polyps and CRC detection

Exclusion Criteria:

-

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals in normal risk for developing CRC aged 50-75 years who undergo preventive colonoscopy for polyps and CRC detection
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Genes' mutations rate in patients who are submitted screening colonoscopy and they presented with no endoscopic findings | 1 month
Genes' mutations rate in patients who are submitted screening colonoscopy and they presented with adenomatous polyp bigger than 1 cm | 1 month
Genes' mutations rate in patients who are submitted screening colonoscopy and they presented with cancerous lesion | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Viazis, Director, Principal Investigator — Evangelismos Hospital
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece

REFERENCES:
- [Result] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Result] Pox CP, Altenhofen L, Brenner H, Theilmeier A, Von Stillfried D, Schmiegel W. Efficacy of a nationwide screening colonoscopy program for colorectal cancer. Gastroenterology. 2012 Jun;142(7):1460-7.e2. doi: 10.1053/j.gastro.2012.03.022. Epub 2012 Mar 21. PMID 22446606
- [Result] Deschoolmeester V, Baay M, Specenier P, Lardon F, Vermorken JB. A review of the most promising biomarkers in colorectal cancer: one step closer to targeted therapy. Oncologist. 2010;15(7):699-731. doi: 10.1634/theoncologist.2010-0025. Epub 2010 Jun 28. PMID 20584808
- [Result] Pino MS, Chung DC. The chromosomal instability pathway in colon cancer. Gastroenterology. 2010 Jun;138(6):2059-72. doi: 10.1053/j.gastro.2009.12.065. PMID 20420946
- [Result] Boland CR, Goel A. Microsatellite instability in colorectal cancer. Gastroenterology. 2010 Jun;138(6):2073-2087.e3. doi: 10.1053/j.gastro.2009.12.064. PMID 20420947
- [Result] Schee K, Fodstad O, Flatmark K. MicroRNAs as biomarkers in colorectal cancer. Am J Pathol. 2010 Oct;177(4):1592-9. doi: 10.2353/ajpath.2010.100024. Epub 2010 Sep 9. PMID 20829435
- [Result] Shen L, Toyota M, Kondo Y, Lin E, Zhang L, Guo Y, Hernandez NS, Chen X, Ahmed S, Konishi K, Hamilton SR, Issa JP. Integrated genetic and epigenetic analysis identifies three different subclasses of colon cancer. Proc Natl Acad Sci U S A. 2007 Nov 20;104(47):18654-9. doi: 10.1073/pnas.0704652104. Epub 2007 Nov 14. PMID 18003927
- [Result] Soreide K, Janssen EA, Soiland H, Korner H, Baak JP. Microsatellite instability in colorectal cancer. Br J Surg. 2006 Apr;93(4):395-406. doi: 10.1002/bjs.5328. PMID 16555243
- [Result] Baylin SB, Hoppener JW, de Bustros A, Steenbergh PH, Lips CJ, Nelkin BD. DNA methylation patterns of the calcitonin gene in human lung cancers and lymphomas. Cancer Res. 1986 Jun;46(6):2917-22. PMID 3009002